CLINICAL TRIAL: NCT06467669
Title: Predictive Outcomes for Selective Thumb Carpometacarpal Joint Denervation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REB24-0025
Record Dates: First submitted 2024-06-07; First posted 2024-06-21 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: CMC Arthritis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participants (Experimental): Patients with 1st CMC arthritis with Eaton stage 2 or 3 disease
  Interventions: Other: Wrist denervation procedure

INTERVENTIONS:
Other: Wrist denervation procedure — To summarize, a Wagner incision is made starting over the junction of the glabrous and non-glabrous skin overlying the thumb CMC joint extending toward the distal wrist crease. The branches of the superficial radial nerve are identified as lying perpendicular to the plane overlying the fascia of the thenar muscles. The branches of the lateral antebrachial cutaneous nerve are identified and resected within the anatomic snuffbox deep to the first compartment. Finally, the thenar muscle fibers are divided at their proximal origin to identify the articular branches of the posterior cutaneous branch of the median nerve.

SUMMARY:
Background: The thumb (or first) carpometacarpal (CMC) joint is commonly affected by osteoarthritis. Literature has reported a prevalence of 15% in women and 7% in men. First CMC joint osteoarthritis can present with decreased grip strength, pain, instability and inability to engage in routine daily activities. Definitive management is with surgery, however these are associated with known risks and increased weight times for the patient. First CMC joint denervation surgery is supported in the literature as a safe and effective approach to treat pain, strength, and thumb opposition which still allows for definitive surgery to be performed later if the arthritis progressed or if the pain returned later after the surgery.

Objectives: (1) evaluate the effectiveness of the neurectomy in patients with with CMC arthritis with respect to pain relief, functional parameters, and Quick disabilities of the arm, shoulder and hand (QuickDASH) scores; (2) to determine whether pain relief with selective nerve blocks are predictive of the outcome of the combined neurectomy; and (3) to determine whether improvement in grip strength following selective blocks is predictive of final grip strength and outcome following neurectomy.

Methods: Patients referred to the plastic surgery clinic for assessment of symptomatic first CMC joint osteoarthritis will be provided options for standard treatment or denervation procedure. Patients who agree to denervation will undergo local anesthetic block at their initial consult. At their initial consultation as well as at the 2-week, 3-month, 6-month, 12-month and 24-month post-surgical follow-up, patients will complete a QuickDASH, Kapandji score, pain scores, 2-point discrimination and grip/key/3-point strength measurements. The total patient population included in this study will be 60 patients.

ELIGIBILITY:
Inclusion Criteria:

* Radiographic Eaton stage 2 or 3 1st carpometacarpal joint arthritis
* Failed medical management, requesting surgical intervention

Exclusion Criteria:

* Pediatric population
* Eaton stage 1 or 4
* Medically unfit for procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Pain outcomes from neurectomy | 2 years
  Participants will have their pre-operative pain scores compared to their post-operative denervation procedure evaluated with a QuickDASH questionnaire. This form will be completed at pre-operative visits and each follow-up appointment.

SECONDARY OUTCOMES:
Selective nerve block pain predictions | 2 years
  Number of participants with changes in pain with pre-operative selective nerve blocks evaluated on the Quick DASH questionnaire will be compared to the scores on the same questionnaire following the denervation procedure at each follow-up visit.
Selective nerve block grip strength predictions | 2 years
  Participants will have grip strength measurements with pre-operative selective nerve blocks evaluated by the key-pinch and 3-point strength tests will be compared to the grip strength measurements at each follow-up visit following the denervation procedure on the same scale.

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Knox, MD, Principal Investigator — University of Calgary

IPD SHARING:
Plan to Share IPD: No
Depending on interest from other Institutions across Canada who wish to participate and make this a nationwide study, we may make a plan for this data to be available to other research teams.

REFERENCES:
- [Result] Haara MM, Heliovaara M, Kroger H, Arokoski JP, Manninen P, Karkkainen A, Knekt P, Impivaara O, Aromaa A. Osteoarthritis in the carpometacarpal joint of the thumb. Prevalence and associations with disability and mortality. J Bone Joint Surg Am. 2004 Jul;86(7):1452-7. doi: 10.2106/00004623-200407000-00013. PMID 15252092
- [Result] Pickrell BB, Eberlin KR. Thumb Basal Joint Arthritis. Clin Plast Surg. 2019 Jul;46(3):407-413. doi: 10.1016/j.cps.2019.02.010. PMID 31103085
- [Result] Raj S, Clay R, Ramji S, Shaunak R, Dadrewalla A, Sinha V, Shaunak S. Trapeziectomy versus joint replacement for first carpometacarpal (CMC 1) joint osteoarthritis: a systematic review and meta-analysis. Eur J Orthop Surg Traumatol. 2022 Aug;32(6):1001-1021. doi: 10.1007/s00590-021-03070-5. Epub 2021 Jul 9. PMID 34244850
- [Result] Wajon A, Vinycomb T, Carr E, Edmunds I, Ada L. Surgery for thumb (trapeziometacarpal joint) osteoarthritis. Cochrane Database Syst Rev. 2015 Feb 23;2015(2):CD004631. doi: 10.1002/14651858.CD004631.pub4. PMID 25702783
- [Result] Clarke S, Hagberg W, Kaufmann RA, Grand A, Wollstein R. Complications with the use of Artelon in thumb CMC joint arthritis. Hand (N Y). 2011 Sep;6(3):282-6. doi: 10.1007/s11552-011-9332-x. Epub 2011 Apr 9. PMID 22942852
- [Result] Tuffaha SH, Quan A, Hashemi S, Parikh P, O'Brien-Coon DM, Broyles JM, Dellon AL, Lifchez SD. Selective Thumb Carpometacarpal Joint Denervation for Painful Arthritis: Clinical Outcomes and Cadaveric Study. J Hand Surg Am. 2019 Jan;44(1):64.e1-64.e8. doi: 10.1016/j.jhsa.2018.04.030. Epub 2018 Jun 20. PMID 29934083
- [Result] Suresh V, Frost CM, Lifchez SD. Selective Thumb Carpometacarpal Joint Denervation for Painful Arthritis: Follow-Up of Long-Term Clinical Outcomes. J Hand Surg Glob Online. 2022 Mar 31;5(1):108-111. doi: 10.1016/j.jhsg.2022.02.005. eCollection 2023 Jan. PMID 36704380
- [Result] Mobargha N, Rein S, Hagert E. Ligamento-Muscular Reflex Patterns Following Stimulation of a Thumb Carpometacarpal Ligament: An Electromyographic Study. J Hand Surg Am. 2019 Mar;44(3):248.e1-248.e9. doi: 10.1016/j.jhsa.2018.06.011. Epub 2018 Aug 26. PMID 30158062
- [Result] Rezzadeh K, Rossi K, Trerotola CC, Shah A. First Carpometacarpal Joint Denervation: A Systematic Review. J Hand Surg Am. 2022 Aug;47(8):793.e1-793.e8. doi: 10.1016/j.jhsa.2021.07.020. Epub 2021 Sep 8. PMID 34509313
- [Result] Hofmeister EP, Moran SL, Shin AY. Anterior and posterior interosseous neurectomy for the treatment of chronic dynamic instability of the wrist. Hand (N Y). 2006 Dec;1(2):63-70. doi: 10.1007/s11552-006-9003-5. PMID 18780027
- [Result] Kennedy CD, Manske MC, Huang JI. Classifications in Brief: The Eaton-Littler Classification of Thumb Carpometacarpal Joint Arthrosis. Clin Orthop Relat Res. 2016 Dec;474(12):2729-2733. doi: 10.1007/s11999-016-4864-6. Epub 2016 May 4. No abstract available. PMID 27146653
- [Result] Kersten P, White PJ, Tennant A. Is the pain visual analogue scale linear and responsive to change? An exploration using Rasch analysis. PLoS One. 2014 Jun 12;9(6):e99485. doi: 10.1371/journal.pone.0099485. eCollection 2014. PMID 24921952
- [Result] Villafane JH, Silva GB, Diaz-Parreno SA, Fernandez-Carnero J. Hypoalgesic and motor effects of kaltenborn mobilization on elderly patients with secondary thumb carpometacarpal osteoarthritis: a randomized controlled trial. J Manipulative Physiol Ther. 2011 Oct;34(8):547-56. doi: 10.1016/j.jmpt.2011.08.005. Epub 2011 Sep 6. PMID 21899891
- [Result] Villafane JH, Cleland JA, Fernandez-de-Las-Penas C. The effectiveness of a manual therapy and exercise protocol in patients with thumb carpometacarpal osteoarthritis: a randomized controlled trial. J Orthop Sports Phys Ther. 2013 Apr;43(4):204-13. doi: 10.2519/jospt.2013.4524. Epub 2013 Mar 13. PMID 23485660
- [Result] Villafane JH, Valdes K, Vanti C, Pillastrini P, Borboni A. Reliability of handgrip strength test in elderly subjects with unilateral thumb carpometacarpal osteoarthritis. Hand (N Y). 2015 Jun;10(2):205-9. doi: 10.1007/s11552-014-9678-y. PMID 26034431